CLINICAL TRIAL: NCT04725669
Title: Seroprevalence of Pertussis Antibodies Among Children and Adolescents in Croatia - Investigation of the Waning Vaccine-induced Immunity in Children and Adolescents
Brief Title: Seroprevalence of Pertussis Among Children and Adolescents in Croatia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital for Infectious Diseases, Croatia (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UHID-06
Record Dates: First submitted 2021-01-20; First posted 2021-01-27 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Immunogenicity, Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Seroprevalence of pertussis among children and adolescents in Croatia (Other): For all patients participating in the study one serum sample will be collected for serological analysis.
  Interventions: Diagnostic Test: ELISA IgG Testkit

INTERVENTIONS:
Diagnostic Test: ELISA IgG Testkit — All samples will be tested for IgG antibody level to pertussis toxin using a commercial Bordetella pertussis ELISA IgG Testkit in accordance to the manufacturers' protocol in the laboratory at the University Hospital for Infectious Diseases in Zagreb.

SUMMARY:
Pertussis is a vaccine preventable disease caused by Bordetella pertussis. Older children and adolescents with pertussis continue to be a significant source of infection for incompletely vaccinated infants who are in harm for developing severe disease. The primary objective of our study is to estimate the duration of protection elicited by the current vaccination schedule against pertussis in Croatia.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents from 6 to 18 years of age treated through Emergency room and/or Day hospital of Pediatric Infectious Diseases Department at UHID;
* appropriate vaccination with pertussis component containing vaccine by date and at the appropriate time, according to Croatian NIP proven by insight in the Vaccination Record Card
* written informed consent obtained from the subject's parent or caregiver, as well as from participants ≥ 16 years old.

Exclusion Criteria:

* children under 6 years
* children and adolescents with acute respiratory symptoms
* children and adolescents with pertussis-like illness within 12 months
* children and adolescents with unknown, uncompleted or irregular vaccination record
* inpatients
* children and adolescents with immunodeficiencies

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1500 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-06-14 (Estimated); Study Completion 2022-09-08 (Estimated)

PRIMARY OUTCOMES:
Waning of vaccine-induced immunity | 1 day
  Number of Participants In Each Specific Age Group With Negative Pertussis Toxin IgG Antibody Titre Measured by ELISA IgG Testkit

SECONDARY OUTCOMES:
Seroprevalence | up to 6 months
  Prevalence of Pertussis Toxin IgG Antibody Titre At Each Specific Age Subgroup

CONTACTS AND LOCATIONS:
Overall Officials: Goran Tešović, Principal Investigator — University Hospital for Infectious Diseases "Dr Fran Mihaljević"
Locations (1):
- University Hospital for Infectious Diseases "Dr Fran Mihaljević", Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No